CLINICAL TRIAL: NCT02089607
Title: Clinical Outcomes and Quality of Life Measures in Patients Treated for Complex Abdominal, Thoracoabdominal and Aortic Arch Aneurysms or Dissections With Fenestrated and Branched Stent Grafts
Brief Title: CAAAs, TAAAs, Aortic Arch Aneurysms or Dissections With Fenestrated/Branched Stent Graft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: William Cook Australia (Industry)
Responsible Party: Principal Investigator, Gustavo S Oderich, Michael E. DeBakey Distinguished Endowed Chair in Surgery, Professor of Surgery, Chief of Division of Vascular Surgery and Endovascular Therapy, Director of Baylor Medicine Center for Aortic Surgery, MICHAEL E. DEBAKEY DEPARTMENT OF SURGERY, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-56531
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Complex Abdominal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm; Aortic Arch Aneurysm; Aortic Arch Dissection
Keywords: aneurysm; aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aneurysm, Aortic Arch; Dissection, Thoracic Aorta; Aneurysm; Aortic Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Complex Abdominal (CAAA) and Thoracoabdominal Aortic Aneurysm (TAAA) Arm (Experimental): The CAAA and TAAA study arm will include 700 patients treated by endovascular aortic repair of CAAAs and TAAAs (Extent I to IV) using either an off-the-shelf Zenith t-Branch or patient-specific stent-graft with a combination of fenestrations and/or branches, with or without concomitant unilateral or bilateral iliac artery aneurysms treated by iliac branch devices. The graft includes 1 to 5 small holes (fenestrations) or cuffs (side branches). These small holes or branches are the investigational part of this research study. The arteries to the liver, intestine, and kidneys will have a stent (small tubular stainless steel structures) to help keep the arteries open and aligned with the fenestrations or branches.
  Interventions: Device: CAAA and TAAA Arm
- Aortic Arch Aneurysm Arm (Experimental): Aortic Arch study arm will include 60 patients with aortic arch aneurysms treated by patient-specific stent-grafts with one to three inner branches or a scallop.
  The study will include patients with CAAAs, TAAAs and/or aortic arch aneurysms due to degenerative aneurysms or chronic aortic dissections. The stent-graft design for this study will be individually selected based on anatomy at the discretion of the principal investigator.
  Interventions: Device: Aortic Arch Aneurysm Arm

INTERVENTIONS:
Device: CAAA and TAAA Arm — The Zenith Fenestrated-Branched System is a tubular graft made of polyester fabric sewn to stainless steel stents that keep the graft open. The graft will be inserted through arteries in the leg (called endovascular repair). This procedure uses catheters that go inside the blood vessel to place a stent graft above and below the aneurysm. The graft includes 1 to 5 small holes (fenestrations) or cuffs (side branches). One or more than one of the study devices including the Zenith® Fenestrated AAA Endovascular Graft, Zenith® t-Branch Endovascular Graft, Patient-Specific Thoracoabdominal Graft, Patient-Specific Distal Bifurcated Component, and Zenith® Branch Endovascular Graft-Iliac Bifurcation will be implanted. The arteries to the liver, intestine, and kidneys will have a stent (small tubular stainless steel structures) to help keep the arteries open and aligned with the fenestrations or branches.
  Other Names: Endovascular stent; Stent-graft
  Arms: Complex Abdominal (CAAA) and Thoracoabdominal Aortic Aneurysm (TAAA) Arm
Device: Aortic Arch Aneurysm Arm — The Zenith® Arch Branch Endovascular Graft includes the main aortic arch portion and one to three cuffs (side branches) that allow the graft to be located in the aortic arch. The number of cuffs is decided based on the anatomy of your aneurysm. The arteries in the aortic arch are the innominate artery (Zone 0), left common carotid artery (Zone 1) and the left subclavian artery (Zone 2). These arteries supply the right arm and right side of the brain, the left side of the brain and the left arm, respectively. The main aortic endovascular graft will be connected into the innominate artery, left common carotid artery and left subclavian artery using additional stents into the branch vessels.
  Arms: Aortic Arch Aneurysm Arm

SUMMARY:
The purpose of this study is to gather safety and effectiveness of the Zenith t-Branch and customized physician-specified stent-graft with a combination of fenestrations and/or branches to repair aortic aneurysm.

DETAILED DESCRIPTION:
This is a traditional device feasibility study intended to generate preliminary safety and efficacy information that may be used to plan an appropriate future study, or to inform further product development.

Subjects will have been diagnosed with a bulge or aneurysm in their aortic arch and or abdominal aorta, which is the blood vessel in the abdomen (belly) that supplies blood to most of the lower body including major organs and the legs.

The Zenith t-Branch and physician-specified fenestrated and branched endovascular graft is a tubular graft made of polyester fabric sewn to stainless steel stents that keep the graft open. As an aneurysm expands, the walls become weak and may rupture, causing a major loss of blood with a high risk of death and other serious complications. To avoid this risk the aneurysm will be repaired by putting a graft inside the aneurysm. The graft will be inserted through arteries in the groin (called endovascular repair). This procedure uses catheters that go inside the blood vessel to place a stent-graft above and below the aneurysm.

The graft includes 1 to 5 small holes (fenestrations) or cuffs (side branches). These small holes or branches are the investigational part of this research study. The arteries to the liver, intestine, and kidneys will have a stent (small tubular stainless steel structures) to help keep the arteries open and aligned with the fenestrations or branches. The Zenith t-Branch and physician-specified fenestrated and branched endovascular graft will be referred to as the Zenith Fenestrated-Branched System.

ELIGIBILITY:
General Inclusion Criteria:

* Thoracoabdominal aortic aneurysm with a diameter ≥ 5.5 cm or 2 times the normal aortic diameter.
* Aneurysm with a history of growth ≥ 0.5 cm per year.
* Saccular aneurysms deemed at significant risk for rupture based upon physician interpretation.
* Presence of concomitant thoracoabdominal and aortic arch aneurysm meeting one of the above-mentioned criteria.
* Presence of thoracoabdominal aortic aneurysm meeting one of the above-mentioned criteria with unilateral or bilateral common iliac artery aneurysm with diameter ≥ 3.0-cm or saccular morphology with no suitable landing zone proximal to iliac bifurcation.

General Exclusion Criteria:

* Less than 18 years of age
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent by the patient or a legally authorized representative
* Pregnant or breastfeeding
* Life expectancy < 2 years
* Prior open surgical or interventional procedure within 30 days of the anticipated date of the fenestrated-branched procedure, with the exception of planned staged procedures to provide access for repair (e.g. staged iliac conduit, cervical debranching, elephant trunk repair), to facilitate the procedure by allowing open revascularization of a target artery not amenable to revascularization with the investigational device, such as an internal iliac artery, subclavian artery or visceral artery with early bifurcation, tortuosity or occlusive disease preventing successful placement of alignment side stents.
* Participation in another investigational clinical or device trial, with the exception of participation in another investigational endovascular stent-graft protocol, percutaneous aortic valve protocol, or concomitant clinical trials designed to evaluate medical therapy strategies to reduce perioperative risk during fenestrated-branched endovascular repair, including risks of renal dysfunction, contrast-induced nephropathy, neurologic, spinal cord or cardiac complications, and/or use of advanced imaging to reduce radiation exposure during implantation of these devices. Participation in investigational device trials not encompassed by the IDE protocol should be performed remotely from the fenestrated procedure (> 30 days). Examples include remote (>30 days) participation in a thoracic, abdominal or iliac branch device trial, or participation in a percutaneous aortic valve trial. Participation in medical therapy trial or advanced imaging trial designed to improve peri-operative outcomes or to reduce radiation exposure of fenestrated-branched endografts may be concurrent with the IDE study. Examples include therapy directed to reduce rates of spinal cord injury, stroke and contrast-induced nephropathy associated with implantation of fenestrated-branched stent-grafts or advanced imaging trials designed to reduce radiation exposure during repair.
* Patients with ruptured aortic aneurysms requiring urgent or emergent repair, with the exception of patients with contained, stable ruptures with anatomy suitable for an off-the-shelf design.

Medical Exclusion Criteria:

* Known sensitivities or allergies to stainless steel, nitinol, polyester, solder (tin, silver), polypropylene, PTFE, urethane or gold
* History of anaphylactic reaction to contrast material that cannot be adequately pre-medicated
* Leaking or ruptured aneurysm associated with hypotension
* Uncorrectable coagulopathy
* Mycotic aneurysm or patients with evidence of active systemic infection.
* History of connective tissue disorder (e.g vascular Ehlers Danlos, Marfans syndrome), with the exception of those patients who had prior open surgical aortic replacement, where a surgical graft would serve as landing zone for the investigational stent-graft, those who are deemed prohibitive risk for open surgical repair or connective tissue disorders with no effect of vascular system (e.g non-vascular forms of Ehlers Danlos).
* Body habitus that would inhibit X-ray visualization of the aorta and its branches.

Anatomical Exclusion Criteria:

* Inadequate femoral or iliac access compatible with the required delivery systems.
* Inability to perform a temporary or permanent open surgical or endovascular iliac conduit for patients with inadequate femoral/iliac access.
* Absence of a non-aneurysmal aortic segment in the distal thoracic aorta above the diaphragmatic hiatus with: a. A diameter measured outer wall to outer wall of no greater than 42mm and no less than 21 mm; b. Parallel aortic wall with <20% diameter change and without significant calcification and/or thrombus in the selected area of seal zone
* Visceral vessel anatomy not compatible with Zenith t-Branch or patient-specific stent-graft due to excessive occlusive disease or small size not amenable to stent graft placement
* Unsuitable distal iliac artery fixation site and anatomy for iliac limb extension or iliac branch device: a. Common iliac artery fixation site diameter, measured outer wall to outer wall on a sectional image (CT) <8.0 mm with inability to perform open surgical conduit ; b. Iliac artery diameter, measured outer wall to outer wall on a sectional image (CT) >20 mm at distal fixation site, with inability to perform open internal iliac artery revascularization or iliac branch stent graft ; c. Non-aneurysmal external liac artery distal fixation site <10 mm in length ; d. Non-aneurysmal internal iliac artery main trunk or branch segment with length <10mm or with inner wall diameter <4 or >14mm; e. Unsuitable anatomy due to inability to preserve at least one hypogastric artery

Additional anatomical inclusion criteria for aortic arch devices:

* Proximal aortic fixation zone: a. Native aorta or surgical graft; b. Diameter: 20-42mm; c. Proximal neck length ≥ 20mm; d. Ascending aortic length ≥50mm; e. Must occur distal to coronary arteries and any coronary artery bypass grafts that are considered patent and necessary for proper cardiac perfusion
* Distal aortic fixation zone:; a. Native aorta or surgical graft; b. Diameter: 20-42mm; c. Distal neck length ≥20mm
* Supra-aortic trunk (brachiocephalic) vessels: a. Although the prosthesis will typically have two branches, modifications to the design will allow for a single branch, three branches or combination of branch and scallop if a customized version is required. Thus, it is generally planned that at least one extra-anatomic bypass graft will be done in conjunction (or in a staged fashion) with the procedure, unless three branches are planned. The two vessels incorporated into the endograft repair would most commonly be the innominate artery and left common carotid artery. However, the innominate artery may be coupled with the left subclavian artery in the setting of a bovine arch whereby the flow to the left carotid would come from a left subclavian to carotid bypass. Similarly, the left carotid and subclavian artery may be branched, or simply one vessel branched should specific anatomic limitations exist. In such a situation, multiple extra-anatomic bypasses may be necessary. A design with a single subclavian retrograde branch and double scallop to the left carotid artery may be used to extent the landing zone to Zone 1. Finally, a design with two antegrade inner branches for the innominate and left common carotid, and one retrograde inner branch for the left subclavian artery may be used in select cases. Thus the inclusion criteria are defined for each artery, yet any combination of arteries may be used for a repair: Innominate artery (Native vessel or surgical graft, Diameter: 8-22mm, Length of sealing zone ≥10mm, Acceptable tortuosity); Left (or right) common carotid artery (Native vessel or surgical graft, Diameter 6-16mm, Length of sealing zone ≥10mm, Acceptable tortuosity); Left (or right) common carotid artery (Native vessel or surgical graft, Diameter: 5-20mm, Length of sealing zone ≥10mm, Acceptable tortuosity).
* In the setting of an aortic dissection the following criteria must exist: a. Access into the true lumen from the groin and at least one supra-aortic trunk vessel; b. A sealing zone in the target aorta (or surgical graft) that is proximal to the primary dissection, such that a stent-graft would be anticipated to seal off the dissection lumen; c. A sealing zone in the target supra-aortic trunk vessels that is distal to the dissection, anticipated to seal off the dissection lumen, or surgically created; d. A true lumen size large enough to deploy the device and still gain access into the target branches
* In the setting of more distal disease: a. The repair may be coupled with a thoracoabdominal branched device, infrarenal device, and/or internal iliac branch device.
* Iliac anatomy must allow for the delivery of the arch branch device which is loaded within a 20F-24F sheath. Thus the iliac requirements are no different than the standard thoracic protocol. Conduits to the iliac vessels or aorta may be used if deemed necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who have died at 30 days post treatment | 30 days post treatment
  Deaths 30 days after treatment
Number of subjects who experience a Major Adverse Event at 30 days post treatment | 30 days post treatment
  A Major Adverse Event includes any of the following: bowel ischemia, myocardial infarction (heart attack), paraplegia, renal failure, respiratory failure, stroke, or blood loss greater than 1000 ml.

SECONDARY OUTCOMES:
Percentage of subjects who achieve treatment success | 12 months post treatment
  Treatment success is defined by a composite endpoint, which includes all the following criteria: 1) technical success, defined as successful delivery and deployment of the custom-made endovascular graft with preservation of those branch vessels intended to be preserved; 2) freedom from type I or III endoleak; 3) freedom from stent-graft migration; 4) freedom from aneurysm enlargement >5 mm; 5) freedom from aneurysm rupture or conversion to open repair.
Mean Quality of Life Measure at Various Time Points | Pre-procedure, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Subjects complete the Short-Form General Health Survey (SF-36) form which consists of an 11 question survey that is divided into 2 parts: physical and emotional. The scale scores range from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo S. Oderich, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chait J, Tenorio ER, Kawajiri H, Lima GBB, Cirillo-Penn NC, Bagameri G, Pochettino A, DeMartino RR, Oderich GS, Mendes BC. Mid-Term Outcomes of "Complete Aortic Repair": Surgical or Endovascular Total Arch Replacement With Thoracoabdominal Fenestrated-Branched Endovascular Aortic Repair. J Endovasc Ther. 2025 Apr;32(2):503-512. doi: 10.1177/15266028231181211. Epub 2023 Jun 14. PMID 37313951
- [Result] Cirillo-Penn NC, MacArthur TA, Tenorio ER, DeMartino RR, Macedo TA, Oderich GS, Mendes BC. Outcomes of patients treated with double-wide scallop vs fenestrations for celiac artery incorporation during repair of complex abdominal aortic aneurysms. J Vasc Surg. 2025 May;81(5):1033-1039. doi: 10.1016/j.jvs.2025.01.194. Epub 2025 Jan 28. PMID 39884565
- [Result] Vacirca A, Mesnard T, Huang Y, Mendes BC, Jakimowicz T, Schneider DB, Haulon S, Sobocinski J, Beck AW, Schanzer A, Farber MA, Timaran C, Kahlberg A, Kolbel T, Gasper WJ, Mees BME, Gargiulo M, Dias NV, Woongchae AL, Sweet MP, Mani K, Eagleton M, Pedro LM, Verhagen H, Yeung KK, Tsilimparis N, Resch T, Bertoglio L, Ferreira E, Khashram M, Sulzer T, Dias-Neto M, Tenorio ER, Kanamori LR, Jama K, Parodi E, Gomes V, Colon JP, Chiesa R, Panuccio G, Schurink GW, Lemmens C, Gallitto E, Faggioli G, Karelis A, Wanhainen A, Habib M, Gouveia E Melo R, Kappe KO, Mariko van Knippenberg SE, Tran B, Crawford S, Panagrosso M, Melloni A, Bonardelli S, Garcia R, Ribeiro T, Gormley S, Maximus S, Oderich GS; International Multicenter Aortic Research Group. Predictors of failure to rescue after fenestrated-branched endovascular aortic repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2025 Jul;82(1):32-42.e3. doi: 10.1016/j.jvs.2025.02.032. Epub 2025 Mar 5. PMID 40054790
- [Result] Ruiter Kanamori L, Tenorio E, Babocs D, Lima GB, Mendes B, Macedo TA, Maximus S, Huang Y, Oderich GS. Clinical outcomes and quality of life measures among 5-year survivors of fenestrated-branched endovascular aortic repair. J Vasc Surg. 2025 Jun;81(6):1254-1265. doi: 10.1016/j.jvs.2025.01.210. Epub 2025 Feb 2. PMID 39904414
- [Result] Rodrigues DVS, Chait J, Cirillo-Penn NC, DeMartino RR, Vierkant RA, Oderich GS, Mendes BC. Trends in hospitalization of patients undergoing endovascular treatment of thoracoabdominal aortic aneurysms based on cerebrospinal fluid drainage strategy. J Vasc Surg. 2024 Oct;80(4):988-995.e1. doi: 10.1016/j.jvs.2024.05.032. Epub 2024 May 19. PMID 38768834
- [Result] Mesnard T, Sulzer TAL, Kanamori LR, Babocs D, Vacirca A, Baghbani-Oskouei A, Savadi S, Tenorio ER, Mirza A, Saqib N, Mendes B, Macedo T, Verhagen HJM, Huang Y, Oderich GS. Aneurysm sac shrinkage at 1 year after fenestrated-branched endovascular aortic repair of complex aortic aneurysms offers mid-term survival advantage. J Vasc Surg. 2024 Oct;80(4):958-967.e3. doi: 10.1016/j.jvs.2024.05.054. Epub 2024 May 31. PMID 38825213
- [Result] Ruiter Kanamori L, Tenorio ER, Babocs D, Savadi S, Baghbani-Oskouei A, Huang Y, Figueroa A, Tanenbaum M, Costa Filho JE, Baig M, Macedo TA, Timaran CH, Oderich GS. Indications, safety, and effectiveness of transcatheter electrosurgical septotomy during endovascular repair of aortic dissections. J Vasc Surg. 2024 Nov;80(5):1396-1406. doi: 10.1016/j.jvs.2024.07.089. Epub 2024 Jul 27. PMID 39074740
- [Result] Huang Y, Colglazier J, Mendes BC, Pochettino A, Kalra M, Greason KL, Tenorio ER, Harmsen WS, Oderich GS. Target Artery Outcomes Following Endovascular versus Open Surgical Repair of Thoracoabdominal Aortic Aneurysms - A Single Center Comparative Study. Ann Surg. 2024 Nov 25. doi: 10.1097/SLA.0000000000006594. Online ahead of print. PMID 39584778
- [Result] Steadman JA, Tenorio ER, Chait J, Vierkant RA, DeMartino RR, Oderich GS, Mendes BC. Preoperative predictors of nonhome discharge after fenestrated-branched endovascular repair of complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2024 Mar;79(3):469-477.e3. doi: 10.1016/j.jvs.2023.11.015. Epub 2023 Nov 11. PMID 37956958
- [Result] Mesnard T, Vacirca A, Baghbani-Oskouei A, Sulzer TAL, Savadi S, Kanamori LR, Tenorio ER, Mirza A, Saqib N, Mendes BC, Huang Y, Oderich GS. Prospective evaluation of upper extremity access and total transfemoral approach during fenestrated and branched endovascular repair. J Vasc Surg. 2024 May;79(5):1013-1023.e3. doi: 10.1016/j.jvs.2023.12.033. Epub 2023 Dec 21. PMID 38141739
- [Result] Tanenbaum MT, Figueroa AV, Kanamori LR, Costa Filho JE, Soto Gonzalez M, Sulzer T, Mesnard T, Huang Y, Baig MS, Oderich GS, Timaran CH. Early experience with patient-specific unibody bifurcated fenestrated-branched devices for complex endovascular aortic aneurysm repair. J Vasc Surg. 2024 Nov;80(5):1361-1370. doi: 10.1016/j.jvs.2024.06.020. Epub 2024 Jun 17. PMID 38897392
- [Result] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Result] Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zettervall SL, Huang Y, Oderich GS; U.S. Fenestrated and Branched Aortic Research Consortium. Effect of bridging stent graft selection for directional branches on target artery outcomes of fenestrated-branched endovascular aortic repair in the United States Aortic Research Consortium. J Vasc Surg. 2023 Jul;78(1):10-28.e3. doi: 10.1016/j.jvs.2023.03.025. Epub 2023 Mar 21. PMID 36948277
- [Result] Sulzer TAL, Macedo TA, Strissel N, Hesley GK, Lekah A, Tallarita T, Dias-Neto M, Huang Y, Tenorio ER, Vacirca A, Mesnard T, Baghbani-Oskouei A, Savadi S, de Bruin JL, Verhagen HJM, Mendes B, Oderich GS. Changes in renal-mesenteric duplex ultrasound velocities after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Nov;78(5):1162-1169.e2. doi: 10.1016/j.jvs.2023.06.106. Epub 2023 Jul 14. PMID 37453587
- [Result] Wong J, Tenorio ER, Lima G, Dias-Neto M, Baghbani-Oskouei A, Mendes B, Kratzberg J, Ocasio L, Macedo TA, Oderich GS. Early Feasibility of Endovascular Repair of Distal Aortic Arch Aneurysms Using Patient-Specific Single Retrograde Left Subclavian Artery Branch Stent Graft. Cardiovasc Intervent Radiol. 2023 Feb;46(2):249-254. doi: 10.1007/s00270-022-03304-x. Epub 2022 Nov 1. PMID 36319711
- [Result] Tenorio ER, Mirza AK, Lima GBB, Marcondes GB, Wong J, Mendes BC, Saqib N, Khan S, Macedo TA, Oderich GS. Characterization of Secondary Interventions After Fenestrated-branched Endovascular Repair of Complex Aortic Aneurysms and Its Effect on Quality of Life and Patient Survival. Ann Surg. 2023 Jul 1;278(1):140-147. doi: 10.1097/SLA.0000000000005454. Epub 2022 Jul 8. PMID 35801701
- [Result] Rogers RT, Lemmens CC, Tenorio ER, Schurink GWH, DeMartino RR, Oderich GS, Mees BME, Mendes BC. Fenestrated/branched endovascular aortic repair using unilateral femoral access in patients with iliac occlusive disease. J Vasc Surg. 2023 Mar;77(3):722-730. doi: 10.1016/j.jvs.2022.10.049. Epub 2022 Nov 11. PMID 36372375
- [Result] Dias-Neto M, Marcondes G, Tenorio ER, Barbosa Lima GB, Baghbani-Oskouei A, Vacirca A, Mendes BC, Saqib N, Mirza AK, Oderich GS. Outcomes of iliofemoral conduits during fenestrated-branched endovascular repair of complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2023 Mar;77(3):712-721.e1. doi: 10.1016/j.jvs.2022.10.050. Epub 2022 Nov 5. PMID 36343871
- [Result] Vacirca A, Wong J, Baghbani-Oskouei A, Tenorio ER, Huang Y, Mirza A, Saqib N, Sulzer T, Mesnard T, Mendes BC, Oderich GS. Outcomes of fenestrated-branched endovascular aortic repair in patients with or without prior history of abdominal endovascular or open surgical repair. J Vasc Surg. 2023 Aug;78(2):278-288.e3. doi: 10.1016/j.jvs.2023.04.001. Epub 2023 Apr 19. PMID 37080442
- [Result] Paajanen P, Karkkainen JM, Tenorio ER, Mendes BC, Oderich GS. Effect of patient frailty status on outcomes of fenestrated-branched endovascular aortic repair for complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2022 Nov;76(5):1170-1179.e2. doi: 10.1016/j.jvs.2022.05.008. Epub 2022 Jun 11. PMID 35697310
- [Result] Dias-Neto M, Tenorio ER, Lima GBB, Baghbani-Oskouei A, Saqib N, Mendes BC, Mirza AK, Oderich GS. Outcomes of low- and standard-profile fenestrated and branched stent grafts for treatment of complex abdominal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2022 Nov;76(5):1160-1169.e1. doi: 10.1016/j.jvs.2022.05.028. Epub 2022 Jul 8. PMID 35810953
- [Result] Chait J, Tenorio ER, Mendes BC, Barbosa Lima GB, Marcondes GB, Wong J, Macedo TA, De Martino RR, Oderich GS. Impact of gap distance between fenestration and aortic wall on target artery instability following fenestrated-branched endovascular aortic repair. J Vasc Surg. 2022 Jul;76(1):79-87.e4. doi: 10.1016/j.jvs.2022.01.135. Epub 2022 Feb 16. PMID 35181519
- [Result] Tenorio ER, Ribeiro MS, Banga PV, Mendes BC, Karkkainen J, DeMartino RR, Hoffman EM, Oderich GS. Prospective Assessment of a Protocol Using Neuromonitoring, Early Limb Reperfusion, and Selective Temporary Aneurysm Sac Perfusion to Prevent Spinal Cord Injury During Fenestrated-branched Endovascular Aortic Repair. Ann Surg. 2022 Dec 1;276(6):e1028-e1034. doi: 10.1097/SLA.0000000000004624. Epub 2021 Jan 7. PMID 33417331
- [Result] Squizzato F, Oderich GS, Tenorio ER, Mendes BC, DeMartino RR. Effect of celiac axis compression on target vessel-related outcomes during fenestrated-branched endovascular aortic repair. J Vasc Surg. 2021 Apr;73(4):1167-1177.e1. doi: 10.1016/j.jvs.2020.07.092. Epub 2020 Aug 27. PMID 32861863
- [Result] Squizzato F, Oderich GS, Balachandran P, Tenorio ER, Mendes BC, De Martino RR. Effect of aortic angulation on the outcomes of fenestrated-branched endovascular aortic repair. J Vasc Surg. 2021 Aug;74(2):372-382.e3. doi: 10.1016/j.jvs.2021.01.027. Epub 2021 Feb 4. PMID 33548434
- [Result] Marcondes GB, Tenorio ER, Baumgardt G, Mendes B, Oderich GS. Evaluation of Safety of Overhead Upper Extremity Positioning During Fenestrated-Branched Endovascular Repair of Thoracoabdominal Aortic Aneurysms. Cardiovasc Intervent Radiol. 2021 Dec;44(12):1895-1902. doi: 10.1007/s00270-021-02992-1. Epub 2021 Oct 27. PMID 34708266
- [Result] Banga P, Oderich GS, Farber M, Reis de Souza L, Tenorio ER, Timaran C, Schneider DB, Baumgardt Barbosa Lima G, Barreira Marcondes G, Timaran D. Impact of Number of Vessels Targeted on Outcomes of Fenestrated-Branched Endovascular Repair for Complex Abdominal Aortic Aneurysms. Ann Vasc Surg. 2021 Apr;72:98-105. doi: 10.1016/j.avsg.2020.09.063. Epub 2020 Nov 21. PMID 33227467
- [Result] Cajas-Monson L, D'Oria M, Tenorio E, Mendes BC, Oderich GS, DeMartino RR. Effect of renal function on patient survival after endovascular thoracoabdominal and pararenal aortic aneurysm repair. J Vasc Surg. 2021 Jul;74(1):13-19. doi: 10.1016/j.jvs.2020.11.040. Epub 2020 Dec 16. PMID 33340697
- [Result] Karkkainen JM, Oderich GS, Tenorio ER, Pather K, Oksala N, Macedo TA, Vrtiska T, Mees B, Jacobs MJ. Psoas muscle area and attenuation are highly predictive of complications and mortality after complex endovascular aortic repair. J Vasc Surg. 2021 Apr;73(4):1178-1188.e1. doi: 10.1016/j.jvs.2020.08.141. Epub 2020 Sep 28. PMID 33002587
- [Result] Oderich GS, Tenorio ER, Mendes BC, Lima GBB, Marcondes GB, Saqib N, Hofer J, Wong J, Macedo TA. Midterm Outcomes of a Prospective, Nonrandomized Study to Evaluate Endovascular Repair of Complex Aortic Aneurysms Using Fenestrated-Branched Endografts. Ann Surg. 2021 Sep 1;274(3):491-499. doi: 10.1097/SLA.0000000000004982. PMID 34132698
- [Result] Karkkainen JM, Tenorio ER, Jain A, Mendes BC, Macedo TA, Pather K, Gloviczki P, Oderich GS. Outcomes of target vessel endoleaks after fenestrated-branched endovascular aortic repair. J Vasc Surg. 2020 Aug;72(2):445-455. doi: 10.1016/j.jvs.2019.09.055. Epub 2020 Jan 21. PMID 31980247
- [Result] Karkkainen JM, Tenorio ER, Pather K, Mendes BC, Macedo TA, Wigham J, Diderrich A, Oderich GS. Outcomes of Small Renal Artery Targets in Patients Treated by Fenestrated-Branched Endovascular Aortic Repair. Eur J Vasc Endovasc Surg. 2020 Jun;59(6):910-917. doi: 10.1016/j.ejvs.2020.02.015. Epub 2020 Mar 18. PMID 32197996
- [Result] Sen I, Tenorio ER, Mirza AK, Karkkainen JM, Mendes BC, DeMartino RR, Cha S, Oderich GS. Effect of Blood Loss and Transfusion Requirements on Clinical Outcomes of Fenestrated-Branched Endovascular Aortic Repair. Cardiovasc Intervent Radiol. 2020 Nov;43(11):1600-1607. doi: 10.1007/s00270-020-02573-8. Epub 2020 Aug 30. PMID 32864718
- [Result] Tenorio ER, Karkkainen JM, Mendes BC, DeMartino RR, Macedo TA, Diderrich A, Hofer J, Oderich GS. Outcomes of directional branches using self-expandable or balloon-expandable stent grafts during endovascular repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2020 May;71(5):1489-1502.e6. doi: 10.1016/j.jvs.2019.07.079. Epub 2019 Oct 11. PMID 31611106
- [Result] Chini J, Mendes BC, Tenorio ER, Ribeiro MS, Sandri GA, Cha S, Hofer J, Oderich GS. Preloaded Catheters and Guide-Wire Systems to Facilitate Catheterization During Fenestrated and Branched Endovascular Aortic Repair. Cardiovasc Intervent Radiol. 2019 Dec;42(12):1678-1686. doi: 10.1007/s00270-019-02322-6. Epub 2019 Aug 27. PMID 31455986
- [Result] Karkkainen JM, Sandri GA, Tenorio ER, Macedo TA, Hofer J, Gloviczki P, Cha S, Oderich GS. Prospective assessment of health-related quality of life after endovascular repair of pararenal and thoracoabdominal aortic aneurysms using fenestrated-branched endografts. J Vasc Surg. 2019 May;69(5):1356-1366.e6. doi: 10.1016/j.jvs.2018.07.060. Epub 2018 Oct 24. PMID 30714570
- [Result] Oderich GS, Ribeiro M, Reis de Souza L, Hofer J, Wigham J, Cha S. Endovascular repair of thoracoabdominal aortic aneurysms using fenestrated and branched endografts. J Thorac Cardiovasc Surg. 2017 Feb;153(2):S32-S41.e7. doi: 10.1016/j.jtcvs.2016.10.008. Epub 2016 Oct 22. PMID 27866781
- [Result] Oderich GS, Ribeiro M, Hofer J, Wigham J, Cha S, Chini J, Macedo TA, Gloviczki P. Prospective, nonrandomized study to evaluate endovascular repair of pararenal and thoracoabdominal aortic aneurysms using fenestrated-branched endografts based on supraceliac sealing zones. J Vasc Surg. 2017 May;65(5):1249-1259.e10. doi: 10.1016/j.jvs.2016.09.038. Epub 2016 Dec 13. PMID 27986479
- [Result] Banga PV, Oderich GS, Reis de Souza L, Hofer J, Cazares Gonzalez ML, Pulido JN, Cha S, Gloviczki P. Neuromonitoring, Cerebrospinal Fluid Drainage, and Selective Use of Iliofemoral Conduits to Minimize Risk of Spinal Cord Injury During Complex Endovascular Aortic Repair. J Endovasc Ther. 2016 Feb;23(1):139-49. doi: 10.1177/1526602815620898. Epub 2015 Dec 4. PMID 26637837
- [Result] Mendes BC, Oderich GS. Endovascular repair of thoracoabdominal aortic aneurysm using the off-the-shelf multibranched t-Branch stent graft. J Vasc Surg. 2016 May;63(5):1394-1399.e2. doi: 10.1016/j.jvs.2016.02.021. PMID 27109801
- [Result] de Souza LR, Oderich GS, Banga PV, Hofer JM, Wigham JR, Cha S, Gloviczki P. Outcomes of total percutaneous endovascular aortic repair for thoracic, fenestrated, and branched endografts. J Vasc Surg. 2015 Dec;62(6):1442-9.e3. doi: 10.1016/j.jvs.2015.07.072. Epub 2015 Sep 12. PMID 26372191